CLINICAL TRIAL: NCT00006041
Title: Vaccination of Patients Who Have Ovarian, Fallopian Tube or Peritoneal Cancer With Glycosylated MUC-1-KLH Conjugate Plus the Immunological Adjuvant QS-21
Brief Title: Vaccine Therapy in Treating Patients With Ovarian, Fallopian Tube, or Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-121; CDR0000068056 (Registry Identifier: PDQ (Physician Data Query)); NCI-H00-0060
Record Dates: First submitted 2000-07-05; First posted 2004-06-28 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — saponin QA-21V1

INTERVENTIONS:
Biological: MUC1-KLH conjugate vaccine
Biological: MUC1-KLH vaccine/QS21
Biological: QS21

SUMMARY:
RATIONALE: Vaccines made from a person's cancer cells may make the body build an immune response to kill the tumor cells.

PURPOSE: Phase I trial to study the effectiveness of vaccine therapy in treating patients who have ovarian, fallopian tube, or peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of immunization with glycosylated MUC-1-KLH vaccine plus adjuvant QS21 in patients with ovarian, fallopian tube, or peritoneal epithelial cancer. II. Determine the dose of this treatment regimen for optimal antibody response in these patients. III. Determine the effect of immunization with this treatment regimen on the T-cell response in these patients.

OUTLINE: This is a dose escalation study of glycosylated MUC-1-KLH vaccine. Patients receive glycosylated MUC-1-KLH vaccine and QS21 subcutaneously once a week on weeks 1-3, 7, and 19. Cohorts of 6 patients receive escalating doses of glycosylated MUC-1-KLH until the dose for optimal antibody response without unacceptable toxicity is determined. Patients are followed at 2 and 12 weeks, and then every 3 months thereafter as long as detectable immunity against MUC-1 persists.

PROJECTED ACCRUAL: A total of 18-24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed ovarian, fallopian tube, or peritoneal epithelial cancer (any stage at diagnosis) Prior cytoreductive surgery required Refractory or recurrent after at least one prior regimen of platinum based chemotherapy No evidence of disease following salvage chemotherapy, defined as: CA125 less than 35 units Negative physical examination No evidence of disease on CT scan of abdomen and pelvis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin, SGOT, and alkaline phosphatase less than 2 times normal Renal: Creatinine less than 1.6 mg/dL Creatinine clearance at least 50 mL/min Other: No other concurrent active invasive malignancy No seafood allergy No positive stool guaiac (excluding hemorrhoids)

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-02; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sabbatini, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States